CLINICAL TRIAL: NCT04476134
Title: The Perioperative Risks of Adverse Events After Cardiac Surgery: a Retrospective Study
Acronym: PRAECS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Du (Other)
Responsible Party: Sponsor-Investigator, Lei Du, professor, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: WestChinaH-2018-01
Record Dates: First submitted 2020-07-13; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Risks of Adverse Events After Cardiac Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with adverse events: patients underwent adverse events after cardiac surgery

SUMMARY:
Cardiac surgeries under cardiopulmonary bypass (CPB) are a major treatment for heart valve disease and coronary artery disease, and over 1-1.25 million such procedures are performed annually worldwide. These procedures are associated with mortality rates of 0.9-4.0% and morbidity rates up to 45.9%.The analysis of perioperative risk factors for these adverse events can provide beneficial help for improving the prognosis of patients undergoing cardiac surgery.Patients undergoing cardiac surgery under CPB at West China Hospital of Sichuan University between January 1, 2011 and June 30, 2017 and the Second Affiliated Hospital in the School of Medicine of Zhejiang University between September 1, 2013 and June 30, 2017 will be enrolled,and demographic data, preoperative and intraoperative data, and postoperative adverse events were collected.Independent perioperative risk factors of death, organ injury and other adverse events in cardiac surgery patients under CPB were studied by univariate and multivariate Logistic regression analysis to provide evidence for prevention and intervention in clinic.

DETAILED DESCRIPTION:
1. Anesthesia management The standard procedures of anesthesia and CPB in the two institutions were applied as described (49, 50). Briefly, anesthesia was induced with midazolam, sufentanil, muscle relaxant and/or etomidate, and maintained by continuous remifentanil infusion and sevoflurane inhalation, combined with intermittent muscle relaxant and sufentanil intravenous injection.
2. CPB management CPB involved a roll pump, a membrane oxygenator, a filter and connecting tubes and was primed with colloid solution of 1000 mL and 500 ml crystalline liquid. During CPB, blood flow was at 2.0-2.4 L/m2/min to maintain mean arterial pressure at 50-80 mmHg. Cold 4:1 blood cardioplegia was used for heart arrest. During CPB, nasopharyngeal temperature was maintained at 32-340C during these procedures and moderate hemodilution was used. All patients received an initial heparin dose of 375 U/kg to achieve systemic anticoagulation, and additional heparin was intermittently injected to maintain activated clotting time longer than 480 s during CPB. After weaning from CPB, heparin was neutralized with protamine in a 1:1 ratio based on the initial heparin dose.
3. Data Collection Form (DCF) In order to minimize the role of potential confounders on adverse outcomes, we will do a systematic search for "risk factor, predictor, adverse outcome, mortality, morbidity, complications, and cardiac surgery" using EMBASE, Cochrane and PubMed databases from Jan 1, 2000 to Dec 31, 2015. All the perioperative potential risk factors mentioned in these studies will be on the DCF.
4. Data collection All variables in the DCF will be retrieved from the Hospital Electronic Medical Record System and medical records. If information on a certain variable cannot be acquired, it will be recorded as ☒. For example, there may be no record of the hemoglobin level on the fifth day after surgery, so we will write ☒ in brackets on the fifth day hemoglobin value.

   After the data collection is finished, the investigators will sign their names on the first page of the DCF.
5. Data Checking Two supervisors will check data promptly. If data are doubted, they will send their questions to the first investigator. According to the Schedule of Events, an "X" will be recorded after the data are confirmed to be correct. Once the whole DCF is completed, the supervisors sign their names and send the DCF to the statisticians.
6. Data Input Data will be input by one statistician using EpiDate3.0 (Odense, Denmark, http://www.epidata.dk/), and another independent statistician will confirm this procedure. Then the CRFs will be stored sequentially.
7. Quality control and quality assurance Diagnosis must be performed strictly according to pre-established definitions. All data in the DCF will be inspected promptly and correctly in order to guarantee reliability. All procedures in this study will be performed by two independent researchers.
8. Statistical analysis Data analysis will be carried out by experienced biostatisticians.Categorical variables are expressed as frequencies (percentages), and compared between patient groups using the chi-squared or Fisher's exact tests. Shapiro-Wilk tests are used to determine the distribution of continuous variables. Normally distributed data are reported as mean ± standard deviation (SD), and compared between groups using one-way ANOVA test. Skewed data are expressed as median [interquartile range (IQR)] and compared between groups using Wilcoxon rank sum tests. The incidence of complications between groups will be performed with the chi-squared test or Fisher's exact tests. Logistic regression analysis will be performed to evaluate risk factors for complications.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Valve replacement or/and coronary artery bypass graft surgery under CPB

Exclusion Criteria:

1. Combined surgery involving ascending aortic replacement surgery or cardiac tumor resection
2. Emergency surgery (defined as surgery performed before the end of the same workday as admission);
3. Died on the operating table, or could not be weaned off CPB;
4. Medical data missing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery under CPB at West China Hospital of Sichuan University between January 1, 2011 and June 30, 2017 and the Second Affiliated Hospital in the School of Medicine of Zhejiang University between September 1, 2013 and June 30, 2017 will be enrolled, because those hospitals launched electronic medical record systems on January 1, 2011 and September 1, 2013, respectively.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
death | up to 30 days
  all-cause death
postoperative complications | up to 30 days
  complications after the cardiac surgery

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
Because this research is ongoing,and individual participant data involve privacy of patients,we have not decided whether sharing data with other researchers.

REFERENCES:
- [Result] Dixon B, Santamaria JD, Reid D, Collins M, Rechnitzer T, Newcomb AE, Nixon I, Yii M, Rosalion A, Campbell DJ. The association of blood transfusion with mortality after cardiac surgery: cause or confounding? (CME). Transfusion. 2013 Jan;53(1):19-27. doi: 10.1111/j.1537-2995.2012.03697.x. Epub 2012 May 11. PMID 22574710
- [Result] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Result] Ghali WA, Ash AS, Hall RE, Moskowitz MA. Statewide quality improvement initiatives and mortality after cardiac surgery. JAMA. 1997 Feb 5;277(5):379-82. PMID 9010169
- [Result] Bridgewater B. Almanac 2012 adult cardiac surgery: the National Society Journals present selected research that has driven recent advances in clinical cardiology. Hellenic J Cardiol. 2013 Jan-Feb;54(1):5-14. PMID 23340123
- [Result] Raiten JM, Ghadimi K, Augoustides JG, Ramakrishna H, Patel PA, Weiss SJ, Gutsche JT. Atrial fibrillation after cardiac surgery: clinical update on mechanisms and prophylactic strategies. J Cardiothorac Vasc Anesth. 2015;29(3):806-16. doi: 10.1053/j.jvca.2015.01.001. No abstract available. PMID 26009291
- [Result] Maganti MD, Rao V, Borger MA, Ivanov J, David TE. Predictors of low cardiac output syndrome after isolated aortic valve surgery. Circulation. 2005 Aug 30;112(9 Suppl):I448-52. doi: 10.1161/CIRCULATIONAHA.104.526087. PMID 16159861
- [Result] Kuitunen A, Vento A, Suojaranta-Ylinen R, Pettila V. Acute renal failure after cardiac surgery: evaluation of the RIFLE classification. Ann Thorac Surg. 2006 Feb;81(2):542-6. doi: 10.1016/j.athoracsur.2005.07.047. PMID 16427848
- [Result] Haase M, Bellomo R, Matalanis G, Calzavacca P, Dragun D, Haase-Fielitz A. A comparison of the RIFLE and Acute Kidney Injury Network classifications for cardiac surgery-associated acute kidney injury: a prospective cohort study. J Thorac Cardiovasc Surg. 2009 Dec;138(6):1370-6. doi: 10.1016/j.jtcvs.2009.07.007. Epub 2009 Sep 5. PMID 19733864
- [Result] McDonagh DL, Berger M, Mathew JP, Graffagnino C, Milano CA, Newman MF. Neurological complications of cardiac surgery. Lancet Neurol. 2014 May;13(5):490-502. doi: 10.1016/S1474-4422(14)70004-3. Epub 2014 Apr 2. PMID 24703207
- [Result] Lomivorotov VV, Efremov SM, Kirov MY, Fominskiy EV, Karaskov AM. Low-Cardiac-Output Syndrome After Cardiac Surgery. J Cardiothorac Vasc Anesth. 2017 Feb;31(1):291-308. doi: 10.1053/j.jvca.2016.05.029. Epub 2016 Jul 29. No abstract available. PMID 27671216
- [Derived] Cheng Z, Wang Y, Liu J, Ming Y, Yao Y, Wu Z, Guo Y, Du L, Yan M. A novel model for predicting a composite outcome of major complications after valve surgery. Front Cardiovasc Med. 2023 May 17;10:1132428. doi: 10.3389/fcvm.2023.1132428. eCollection 2023. PMID 37265563